CLINICAL TRIAL: NCT05750082
Title: Automated Plaque Characterization and Functional Analysis of Coronary CTA Based on OCT Images Using Artificial Intelligence
Brief Title: The AIPLAQUE Study: An Artificial Intelligence-based Prospective Study to Analyze PLAQUE Using CCTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yu Bo, Director of Department of Cardiology, Harbin Medical University
Other Study IDs: KY2021-003
Record Dates: First submitted 2022-11-08; First posted 2023-03-01 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease Acute Coronary Syndrome Myocardial Ischemia Plaque Characterization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CCTA CT-FR CAG OCT — Per the protocol, patients will have a CCTA (coronary computed tomography angiography), CT-FFR (fractional flow reserve derived from CTA), ICA (invasive coronary angiography), OCT (optical coherence tomography).

SUMMARY:
This trial is a single-center, prospective, observational clinical study. All patients who have at least one coronary artery stenosis of 30%-90% in diameter ≥ 2mm confirmed by CCTA, and who are scheduled to undergo clinically indicated invasive coronary angiography (ICA) and optical coherence tomography (OCT) evaluation and/or treatment will be eligible for enrollment. We proposed a novel approach that integrates CCTA, ICA and OCT images to automatically measure plaque characterization and calculate CT-FFR using computational fluid dynamics (CFD) simulation and artificial intelligence deep learning.

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) is one of the leading causes of coronary artery disease (CAD) death worldwide. Vulnerable plaque rupture is a primary underlying cause of luminal thrombosis responsible for provoking ACS. Therefore, identifying high-risk plaques before ACS occurs has been a major research goal and requires further clinical perspectives. Coronary computed tomography angiography (CCTA) is a comprehensive, non-invasive and cost-effective imaging assessment approach, which can provide the ability to identify the characteristics and morphology of high-risk atherosclerotic plaques associated with ACS. Optical coherence tomography (OCT) is a new, light-based, intravascular imaging technique that provides high-resolution, cross-sectional images of coronary artery anatomy. Due to its superior resolution, OCT is more accurate in measuring the sites of plaque vulnerability, distinguishing the differences in its composition, informing about the anatomic severity of epicardial stenoses, and also provides input for computational models to assess functional severity.

The objectives of the study are: (1) To construct an artificial intelligence model for identifying coronary plaque components on CTA images using OCT as the reference standard. (2) To conduct fluid mechanics simulation including blood vessel wall and plaque by using geometric and physiological models of blood vessels and plaques, and to provide more accurate functional parameters (CT-FFR).

The enrollment criteria will be (1) Patients who presented with stable angina pectoris or acute coronary syndrome; (2) patients who meet the indications for coronary CT angiography, percutaneous coronary angiography and intravascular imaging; (3) Among those patients, patients who have at least one coronary artery stenosis of 30% - 90% in diameter ≥ 2mm confirmed by CCTA.

Data collected will include CCTA, full angiographic, and OCT images. Combined with CTA/ICA/OCT images of multiple modalities, this study will develop a novel images analysis technology to automatically extract vascular lumen, plaque characterization, fluid-solid mechanical properties, and myocardial ischemia conditions using computational fluid dynamics (CFD) simulation and artificial intelligence deep learning.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and able to understand the purpose of the study and sign the informed consent;
2. Patients who presented with stable angina pectoris or acute coronary syndrome;
3. Patients who meet the indications for coronary CT angiography, percutaneous coronary angiography and intravascular imaging;
4. Among those patients, patients who have at least one coronary artery stenosis of 30% - 90% in diameter ≥ 2mm confirmed by CCTA.

Exclusion Criteria:

1. Known pregnancy or breastfeeding at the time of enrollment;
2. Hemodynamic instability;
3. Allergy to contrast media or aspirin, adenosine etc.;
4. History of stroke or transient ischemic attack (TIA) within 12 months before surgery;
5. Known renal insufficiency (e.g. serum creatinine >2.0mg/dL, or creatinine clearance ≤30 mL/min), or need for dialysis, or acute kidney failure (as per physician judgment);
6. Leukopenia (WBC<4.0*10*9/L), thrombocytopenia (PLT<100*10*9/L) or thrombocytopenia (PLT>300*10*9/L);
7. Subjects who receiving oral or intravenous immunosuppressant therapy (other than inhaled steroids) or have an autoimmune disease (e.g., AIDS, SLE; except diabetes);
8. Any other factors that researchers consider not suitable for inclusion or completion of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprised 100 stable patients with angina pectoris or acute coronary syndrome who will receive CCTA, CT-FFR, ICA, and OCT.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
By taking OCT results as the standard, evaluating the accuracy of automated plaque characterization and functional significance of coronary stenosis using CTA images computation. | Immediately after OCT scan
  By taking OCT results as the standard, evaluating the accuracy of automated plaque characterization and functional significance of coronary stenosis using CTA images computation.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China